CLINICAL TRIAL: NCT02415244
Title: Transesophageal Echocardiography (TEE): A Novel Technique for Spinal Cord Imaging
Status: Completed | Type: Observational
Sponsor: Kenichi Ueda (Other)
Responsible Party: Sponsor-Investigator, Kenichi Ueda, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201206753
Record Dates: First submitted 2015-04-08; First posted 2015-04-14 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Spinal Cord; Epidural
Keywords: ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Age 0 - 18: TEE visualization of the spinal cords in patients age between 0 - 18
  Interventions: Procedure: TEE
- Age 18 plus: TEE visualization of the spinal cords in patients age 18 or greater
  Interventions: Procedure: TEE

INTERVENTIONS:
Procedure: TEE — Spinal cord segments will be imaged using the TEE

SUMMARY:
The aim of this prospective observational study is to assess whether transesophageal echocardiography (TEE) can be used to identify the structures within the vertebral foramen of the spinal column and to determine the range of spinal segments which can be visualized.

DETAILED DESCRIPTION:
The aim of this prospective observational study is to assess whether transesophageal echocardiography (TEE) can be used to identify the structures within the vertebral foramen of the spinal column and to determine the range of spinal segments which can be visualized. Data will be collected from both pediatric and adult patients undergoing cardiothoracic and interventional cardiac surgeries under general anesthesia. Because use of TEE is a standard surgical procedure and because TEE will already be in place to visualize the heart, no additional processes will be required to collect data, minimizing patient risk. TEE will be monitored and controlled by a trained anesthesiologist or TEE technician and visualization of the spinal cord will be confirmed. Real-time TEE images will then be captured and later graded by a trained sonographer as high, medium or low quality. Starting at the level of the tracheal bifurcation, corresponding to thoracic vertebral level T5 (Mirajalili 2012), the TEE probe will be advanced cranially to determine the spinal levels visualized above T5 and caudally in order to determine the spinal levels below T5 that can be seen on TEE. At each level seen on TEE, pictures will be taken for confirmation.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for cardiothoracic or interventional cardiac surgeries under general anesthesia

Exclusion Criteria:

* We will exclude any patients with known esophageal abnormalities, lesions or disease that would disqualify the patient for the use of TEE as standard procedure.
* We will also exclude any patients that come to the catheter laboratory exclusively for TEE exam as our study will only occur in patients already scheduled to undergo TEE use in surgery or diagnostic procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All age population going under cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2012-07; Primary Completion 2017-09-23 (Actual); Study Completion 2017-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Ueda, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hosptials and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Background] Pissarra F, Oliveira A, Marcelino P. Transoesophageal echocardiography for monitoring liver surgery: data from a pilot study. Cardiol Res Pract. 2012;2012:723418. doi: 10.1155/2012/723418. Epub 2012 Apr 30. PMID 22611514
- [Background] Chitilian HV, Alston TA, Avery EG. Transesophageal echocardiographic bull's eye. J Cardiothorac Vasc Anesth. 2006 Dec;20(6):894-5. doi: 10.1053/j.jvca.2005.09.007. Epub 2006 Feb 7. No abstract available. PMID 17138103
- [Background] Daniel WG, Erbel R, Kasper W, Visser CA, Engberding R, Sutherland GR, Grube E, Hanrath P, Maisch B, Dennig K, et al. Safety of transesophageal echocardiography. A multicenter survey of 10,419 examinations. Circulation. 1991 Mar;83(3):817-21. doi: 10.1161/01.cir.83.3.817. PMID 1999032
- [Background] Godet G, Couture P, Ionanidis G, Gosgnach M, Kieffer E, Viars P. Another application of two-dimensional transesophageal echocardiography: spinal cord imaging. A preliminary report. J Cardiothorac Vasc Anesth. 1994 Feb;8(1):14-8. doi: 10.1016/1053-0770(94)90005-1. PMID 8167278

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Age 0 - 18 | Age 18 Plus
Started | 50 | 25
Completed | 50 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Age 0 - 18: TEE visualization of the spinal cords in patients age between 0 - 3
  TEE: Spinal cord segments will be imaged using the TEE
- Total: Total of all reporting groups
Arm/Group | Age 0 - 18 | Age 18 Plus | Total
Number analyzed (Participants) | 50 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 0 | 50
  Between 18 and 65 years | 0 | 19 | 19
  >=65 years | 0 | 6 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.0 (4.8) | 52 (20) | 20 (25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 9 | 32
  Male | 27 | 16 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Thoracic Spinal Segments Successfully Visualized With TEE
Description: Count the number of short axis views of thoracic spinal cord segment and surrounding structure visualized with TEE in pediatric and adults patients.
Time Frame: within 30 minutes
Measure: Median (Inter-Quartile Range); unit: Thoracic segments
Groups:
- Pediatric Group: Visible thoracic epidural segments were counted in pediatric patients with TEE
- Adult Group: Visible thoracic epidural segments were counted with TEE
Arm/Group | Pediatric Group | Adult Group
Number analyzed (Participants) | 50 | 25
Thoracic segments | 12 [12 to 12] | 10 [6 to 12]

ADVERSE EVENTS:
Time Frame: within 24 hours
Groups:
- Pediatric Group: Pediatric subjects
- Adult Group: Adult subjects
Arm/Group | Pediatric Group | Adult Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/25
Other Adverse Events (participants affected / at risk) | 0/50 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT02415244/Prot_SAP_001.pdf